CLINICAL TRIAL: NCT01819857
Title: The Influence of Droperidol on Cardiac Repolarization. A Double-blind, Ondansetron-controlled Study.
Brief Title: Droperidol and Cardiac Repolarization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radoslaw Owczuk, Principle Investigator, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RO4; MUG4 (Other: Medical University of Gdansk)
Record Dates: First submitted 2013-03-09; First posted 2013-03-28 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Cardiac Repolarization
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Droperidol 0.625 mg intravenously (Active Comparator)
  Interventions: Drug: Xomolix 0.625 mg intravenously
- Droperidol 1.25 mg intravenously (Active Comparator)
  Interventions: Drug: Xomolix 1.25 mg
- Ondansetron 8 mg intravenously (Active Comparator)
  Interventions: Drug: Zofran 8 mg

INTERVENTIONS:
Drug: Xomolix 0.625 mg intravenously — intravenous administration of 0.625 mg droperidol
  Arms: Droperidol 0.625 mg intravenously
Drug: Xomolix 1.25 mg — intravenous administration of 1.25 mg droperidol
  Arms: Droperidol 1.25 mg intravenously
Drug: Zofran 8 mg — intravenous administration of 8 mg ondansetron
  Arms: Ondansetron 8 mg intravenously

SUMMARY:
For many years droperidol has been used in prophylaxis and therapy of PONV. Information that it can provoke disorders of cardiac ventricular rhythm reduced its popularity. However those data didn't base on solid examinations confirming torsadogenic action of droperidol. It is known that droperidol prolongs time of repolarisation, but there wasn't any data confirming its impact on transmural dispersion of repolarisation. Only estimation both of those actions in one time allows to define for sure arrhythmogenic role of droperidol.

The aim of this study was to answer the questions:

6. Does droperidol make an significant prolongation of heart repolarisation, expressed as corrected QT interval?

1. Does droperidol cause increase of transmural dispersion of repolarisation?
2. Does possible torsadogenic acting of droperidol depend on dose of drug?
3. Does ondansetron cause changes of electrical heart function, suggesting its possibilities to induce TdP tachycardia?
4. What is torsadogenic potential of droperidol and ondansetron used in prophylaxis PONV in people not suffering from cardiovascular diseases?

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* sex: males
* ASA score I or II

Exclusion Criteria:

* treatment with drugs influencing cardiac repolarization
* coronary artery disease
* heart insufficiency NYHA>1
* serum electrolyte disturbances
* hypersensitivity to droperidol and/or ondansetron

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in QT interval value, QTc interval value and transmural dispersion of repolarization (TDR) value | 20 minutes

SECONDARY OUTCOMES:
Number of individuals with QTc increase by 50 ms and TDR increase by 25 ms | 20 min

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdansk, Gdansk, Poland